CLINICAL TRIAL: NCT06330545
Title: A Prospective Clinical Trial of Radiation Therapy for Dupuytren's Contracture Following Surgical and Non-Surgical Release
Brief Title: Radiation Therapy for Dupuytren's Contracture Following Non-Surgical Release
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Lance G. Warhold, Staff Physican, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY02002161
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Dupuytren Contracture
Keywords: Dupuytren's contracture; radiation therapy
MeSH Terms: conditions — Dupuytren Contracture | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: This is a prospective phase II trial where patients diagnosed with late/advanced stage Dupuytren's Contracture (DC) who undergo successful CCH injection and release will receive a standardized regimen of radiotherapy (RT). The study will be powered to assess the outcome in patients undergoing the combination of successful release followed by RT. Patients will be monitored for acute and late toxicities while we evaluate disease recurrence defined as a > 20 degree worsening of contracture in the presence of a palpable cord, or the need for medical/surgical intervention to correct the new or worsening contracture.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Dupuytren's Contacture (Experimental): Patients with Dupuytren's Contacture will undergo Collagenase Clostridium Histolyticum injection and release followed by two 5-day courses of radiation therapy separated by 6-8 weeks. They will then be followed for 3 years for recurrence.
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Patients with Dupuytren's Contacture will undergo Collagenase Clostridium Histolyticum injection and release followed by two 5-day courses of radiation therapy separated by 6-8 weeks. They will then be followed for 3 years for recurrence.

SUMMARY:
The goal of this study is to learn about preventing recurrence of Dupuytren's Contracture. The main question it aims to answer are:

• Does targeted radiation therapy decrease recurrence of Dupuytren's contracture after treatment with Collagenase Clostridium Histolyticum?

Participants will undergo:

* Release of Dupuytren's Contracture after Collagenase Clostridium Histolyticum injection
* Daily radiation therapy treatment for 5 days followed by 6-8 week rest period and then another course of 5 days of radiation therapy

DETAILED DESCRIPTION:
This is a prospective phase II trial where patients diagnosed with late/advanced stage Dupuytren's Contracture (DC) who undergo successful Collagenase Clostridium Histolyticum (CCH) injection and release will receive a standardized regimen of adjuvant radiotherapy (RT). The study will be powered to assess the outcome in patients undergoing the combination of successful release followed by RT. Patients will be monitored for acute and late toxicities while we evaluate disease recurrence defined as a > 20 degree worsening of contracture in the presence of a palpable cord as compared to within 14 days from CCH injection, or the need for medical/surgical intervention to correct the new or worsening contracture.

ELIGIBILITY:
Inclusion Criteria:

* Age 45 or greater with DC
* Extension deficit >10 degrees
* Unable to simultaneously place the affected finger and palm flat on a table.
* Women included in the study will be post-menopausal or using contraception, and a pregnancy test will be performed as standard of care.
* For patients who are having multiple CCH injections, only the first 2 joints on given hand will be included

Exclusion Criteria:

* Unsuccessful non-surgical release (> N/1 disease)
* They develop an open wound during CCH
* Breast feeding or pregnancy
* A chronic muscular, neurologic, or neuromuscular disorder affecting the hands.
* Less than the age of 45
* They have previously undergone radiation on the hand in which they plan to get CCH injections
* They are pregnant women, impaired adults or prisoners

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2032-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence of Dupuytren's Contracture | one month, 6 months, 12 months, 24 months, and 36 months post-radiation treatment
  Recurrence defined as > 20 degrees worsening of contracture relative to within 14 days from CCH injection or the need for medical/surgical intervention to correct the new or worsening symptomatic contracture.
  The investigators will measure the contracture using the table top test in which patients their press hand with best of their ability. We will use a goniometer on dorsal surface of hand while performing table top test to measure PIP and MCP joints.

SECONDARY OUTCOMES:
Radiation Toxicity | one month, 6 months, 12 months, 24 months, and 36 months post-radiation treatment
  acute (30 days or less) and late (> 30 days) Grade 2 and Grade 3 toxicities from radiotherapy defined by Radiation Therapy Oncology Group
Patient Reported Outcomes after Radiation Treatment (RT) | Before Radiation Treatment (RT), after completion of RT, 1-month post-RT, 6 months post-RT, 1 year post-RT, 2 years post-RT, and 3 years post-RT
  The investigators will also record hand function change from baseline to after therapy via the Brief Michigan Hand Questionnaire, a patient reported outcome measure. This questionnaire will be used before study enrollment, after completion of RT, one-month post-RT, six months post-RT, one year post-RT, two years post-RT, and three years post-RT. The Michigan Hand Questionnaire is scored from 0-100 with higher scores indicating better functioning and satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Lance Warhold, MD, Principal Investigator — Dartmouth Health
Locations (1):
- Dartmouth Hitchcock, Lebanon, New Hampshire, United States